CLINICAL TRIAL: NCT05030103
Title: An Open, Prospective Clinical Trial on the Use of Reading Glasses in Children to Prevent Myopia
Brief Title: Myopia Prevention With Reading Glasses
Acronym: SMART2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reis Augenklinik AG (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMART2
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Myopia
Keywords: Children, prevention
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Open, propensity score method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glasses (Active Comparator): The participants are asked to wear reading glasses during near-work. The reading glasses have a lenspower of +2.0 diopters.
  Interventions: Device: Reading glasses, +2.0 diopters
- Control (No Intervention): Age matched children and adolescents, no intervention.

INTERVENTIONS:
Device: Reading glasses, +2.0 diopters — The participants in the glasses-group are asked to wear the reading glasses during near-work.
  Arms: Glasses

SUMMARY:
The last decades have seen a significant increase in myopia in children and young adults. Possible cause: increased near-work (school, computer, smartphone). Rationale: Reading glasses support the accommodative effort of the eyes. By wearing reading glasses, there is less interference with the young eye´s physiological axial growth despite increased near-work. Main objective: does the use of reading glasses during near-work in children and adolescents reduce the incidence of myopia.

DETAILED DESCRIPTION:
In myopia (nearsightedness), the eyeball is relatively to long, which means that the image produced by the cornea and lens is displayed in front of the retina.

The axial length of an adult eye is on average around 23 millimeters. Every millimeter of additional length must be corrected with a -2.75 diopter lens.

In newborns, the eyeball is about 18 millimeters long. It is believed that there are feedback loops during childhood and adolescence to control the growth of the eye.

Epidemiological studies show that myopia is an increasing health problem. There is a growing body of epidemiological evidence that environmental factors can influence the development of myopia.

The link between the environment and myopia lies in the quality of the retinal image. Experimental studies in various species have shown that if the retinal image is missing, eye growth is disturbed. Of even greater importance for the development of myopia is the knowledge that the primate eye can change its growth, depending on the strength and type of blurring of the retinal image: if lenses are placed in front of the eye during development, the eye growth changes in such a way that a sharp retinal image is achieved through these lenses. If divergent lenses are placed in front of the eye, the eye becomes longer, and if convergent lenses are placed in front of it, it becomes correspondingly shorter.

So myopia is the result of a failure in these emmetropization mechanisms. The positive correlation of myopia with a higher level of education suggests that increased close work interferes with emmetropization. The growth in length of the eye changes in such a way that it adapts to this requirement: the eye adjusts itself to the close work: it becomes myopic.

Myopia is thus possibly a physiological adaptation to increased near work with the aim of improving the quality of the retinal image during close work. However, this can only be achieved at the expense of the image quality when looking into the distance.

The investigators submitted a study on this subject to the Cantonal Ethics Committee of the Canton of Zurich in 2003:

"An open, prospective, randomized study on the use of reading glasses in children with normal vision to prevent myopia" Unique Protocol ID: FR-2005-01-01 Approval Status: Approved Approval Number: KEK-StV-Nr. 19/03

This was and is so far the only clinical study that examined the effect of reading glasses on the development of myopia in emmetropic (normally sighted) children and has led to Patent No: US 8,511,819 B2, Aug. 20, 2013 "Prevention of myopia acquisition in children and young adults using reading glasses"

ELIGIBILITY:
Inclusion Criteria:

1. Children of both sexes from the age of 6
2. Children whose parents have read and signed the declaration of consent
3. Spherical equivalent of refraction <-0.5 dpt.
4. Distant vision in both eyes without correction 1.0
5. Willingness to wear reading glasses
6. Possibility of a five-year follow-up

Exclusion Criteria:

1. Children who already wear glasses
2. Astigmatism over 1.5 diopters
3. Anisometropy greater than 1.5 diopters
4. Eye diseases that affect refraction development

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2031-09-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of myopia | Five years
  Number of participants which develop myopia within the follow-up period of five years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Reis, Prof. Dr., Principal Investigator — Reis Augenklinik AG
Locations (1):
- Reis Augenklinik AG, Bendern, Liechtenstein

IPD SHARING:
Plan to Share IPD: No